CLINICAL TRIAL: NCT02305277
Title: Relative Bioavailability and Bioequivalence Of Different Formulations of Opicapone in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-91067-119
Record Dates: First submitted 2014-11-28; First posted 2014-12-02 (Estimated); Results first posted 2015-11-17 (Estimated); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Parkinson
MeSH Terms: interventions — opicapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- BIA 9-1067 5 mg Sequence 1 (Experimental): volunteers received a single oral dose of 5 mg BIA 9-1067: Period 1: CM Formulation Period 2: TBM Formulation
  CM - clinical micronized TBM - to-be-marketed
  Interventions: Drug: BIA 9-1067 (clinical micronized, CM); Drug: BIA 9-1067 (to-be-marketed, TBM)
- BIA 9-1067 25 mg Sequence 1 (Experimental): volunteers received a single oral dose of 25 mg BIA 9-1067: Period 1: CM Formulation Period 2: TBM Formulation
  CM - clinical micronized TBM - to-be-marketed
  Interventions: Drug: BIA 9-1067 (clinical micronized, CM); Drug: BIA 9-1067 (to-be-marketed, TBM)
- BIA 9-1067 50 mg Sequence 1 (Experimental): volunteers received a single oral dose of 50 mg BIA 9-1067: Period 1: CM Formulation Period 2: TBM Formulation
  CM - clinical micronized TBM - to-be-marketed
  Interventions: Drug: BIA 9-1067 (clinical micronized, CM); Drug: BIA 9-1067 (to-be-marketed, TBM)
- BIA 9-1067 5 mg Sequence 2 (Experimental): volunteers received a single oral dose of 5 mg BIA 9-1067: Period 1: TBM Formulation Period 2: CM Formulation
  CM - clinical micronized TBM - to-be-marketed
  Interventions: Drug: BIA 9-1067 (clinical micronized, CM); Drug: BIA 9-1067 (to-be-marketed, TBM)
- BIA 9-1067 25 mg Sequence 2 (Experimental): volunteers received a single oral dose of 25 mg BIA 9-1067: Period 1: TBM Formulation Period 2: CM Formulation
  CM - clinical micronized TBM - to-be-marketed
  Interventions: Drug: BIA 9-1067 (clinical micronized, CM); Drug: BIA 9-1067 (to-be-marketed, TBM)
- BIA 9-1067 50 mg Sequence 2 (Experimental): volunteers received a single oral dose of 50 mg BIA 9-1067: Period 1: TBM Formulation Period 2: CM Formulation
  CM - clinical micronized TBM - to-be-marketed
  Interventions: Drug: BIA 9-1067 (clinical micronized, CM); Drug: BIA 9-1067 (to-be-marketed, TBM)

INTERVENTIONS:
Drug: BIA 9-1067 (clinical micronized, CM)
  Other Names: OPC, Opicapone
Drug: BIA 9-1067 (to-be-marketed, TBM)
  Other Names: OPC, Opicapone

SUMMARY:
Single-centre, open-label, randomised, three-part, two-way crossover study in 84 healthy volunteers. In each part, the study consisted of two consecutive single-dose treatment periods separated by a washout period of at least 14 days.

ELIGIBILITY:
Inclusion Criteria:

* A signed and dated informed consent form before any study-specific screening procedure was performed;
* Male or female subjects aged 18 to 45 years, inclusive;
* Body mass index (BMI) between 18 and 30 kg/m2 inclusive;
* Healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead electrocardiogram (ECG);
* Negative tests for hepatitis B surface antigen (HBsAg), anti- hepatitis C virus antibodies (HCV Ab) and anti-human immunodeficiency virus antibodies (HIV-1 and HIV-2 Ab) at screening;
* Clinical laboratory test results clinically acceptable at screening and admission to each treatment period;
* Negative screen for alcohol and drugs of abuse at screening and admission to each treatment period;
* Non-smokers or ex-smokers for at least 3 months;
* Able to participate, and willing to give written informed consent and comply with the study restrictions.
* If female:
* She was not of childbearing potential by reason of surgery or, if of childbearing potential, she used an effective non-hormonal method of contraception [intrauterine device or intrauterine system; condom or occlusive cap (diaphragm or cervical or vault caps) with spermicidal foam or gel or film or cream or suppository; true abstinence; or vasectomized male partner, provided that he was the sole partner of that subject] for all the duration of the study;
* She had a negative serum pregnancy test at screening and a negative urine pregnancy test at admission to each treatment period.

Exclusion Criteria:

* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders, or had a clinically relevant surgical history;
* Had clinically relevant findings in laboratory tests, particularly any abnormality in the coagulation tests, or any abnormality in the liver function tests;
* Had a history of relevant atopy or drug hypersensitivity;
* Had a history of alcoholism and/or drug abuse;
* Consumed more than 14 units of alcohol per week [1 unit of alcohol = 280 mL beer (3-4°) = 100 mL wine (10-12°) = 30 mL spirits (40°)];
* Had a significant infection or known inflammatory process on screening or admission to each treatment period;
* Had acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission to each treatment period;
* Had used medicines within 2 weeks of admission to first period that could affect the safety or other study assessments, in the Investigator's opinion;
* Had previously received opicapone;
* Had used any investigational drug or participated in any clinical trial within 90 days prior to screening;
* Had participated in more than 2 clinical trials within the 12 months prior to screening;
* Had donated or received any blood or blood products within the 3 months prior to screening;
* Were vegetarians, vegans or had medical dietary restrictions;
* Could not communicate reliably with the Investigator;
* Were unlikely to co-operate with the requirements of the study;
* Were unwilling or unable to give written informed consent;

If female:

* She was pregnant or breast-feeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- BIA 9-1067 5 mg Sequence 1: volunteers received a single oral dose of 5 mg BIA 9-1067: Period 1: CM Formulation Period 2: TBM Formulation
  CM - clinical micronized TBM - to-be-marketed
  BIA 9-1067 (clinical micronized, CM)
  BIA 9-1067 (to-be-marketed, TBM)
- BIA 9-1067 25 mg Sequence 1: volunteers received a single oral dose of 25 mg BIA 9-1067: Period 1: CM Formulation Period 2: TBM Formulation
  CM - clinical micronized TBM - to-be-marketed
  BIA 9-1067 (clinical micronized, CM)
  BIA 9-1067 (to-be-marketed, TBM)
- BIA 9-1067 50 mg Sequence 1: volunteers received a single oral dose of 50 mg BIA 9-1067: Period 1: CM Formulation Period 2: TBM Formulation
  CM - clinical micronized TBM - to-be-marketed
  BIA 9-1067 (clinical micronized, CM)
  BIA 9-1067 (to-be-marketed, TBM)
- BIA 9-1067 5 mg Sequence 2: volunteers received a single oral dose of 5 mg BIA 9-1067: Period 1: TBM Formulation Period 2: CM Formulation
  CM - clinical micronized TBM - to-be-marketed
  BIA 9-1067 (clinical micronized, CM)
  BIA 9-1067 (to-be-marketed, TBM)
- BIA 9-1067 25 mg Sequence 2: volunteers received a single oral dose of 25 mg BIA 9-1067: Period 1: TBM Formulation Period 2: CM Formulation
  CM - clinical micronized TBM - to-be-marketed
  BIA 9-1067 (clinical micronized, CM)
  BIA 9-1067 (to-be-marketed, TBM)
- BIA 9-1067 50 mg Sequence 2: volunteers received a single oral dose of 50 mg BIA 9-1067: Period 1: TBM Formulation Period 2: CM Formulation
  CM - clinical micronized TBM - to-be-marketed
  BIA 9-1067 (clinical micronized, CM)
  BIA 9-1067 (to-be-marketed, TBM)
Period: Overall Study
Arm/Group | BIA 9-1067 5 mg Sequence 1 | BIA 9-1067 25 mg Sequence 1 | BIA 9-1067 50 mg Sequence 1 | BIA 9-1067 5 mg Sequence 2 | BIA 9-1067 25 mg Sequence 2 | BIA 9-1067 50 mg Sequence 2
Started | 15 | 14 | 14 | 14 | 14 | 14
Received CM | 15 | 14 | 14 | 14 | 14 | 14
Received TBM | 15 | 14 | 14 | 14 | 14 | 14
Completed | 14 | 14 | 14 | 14 | 13 | 14
Not Completed | 1 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BIA 9-1067 5 mg Sequence 1 | BIA 9-1067 25 mg Sequence 1 | BIA 9-1067 50 mg Sequence 1 | BIA 9-1067 5 mg Sequence 2 | BIA 9-1067 25 mg Sequence 2 | BIA 9-1067 50 mg Sequence 2 | Total
Number analyzed (Participants) | 15 | 14 | 14 | 14 | 14 | 14 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 14 | 14 | 14 | 14 | 85
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 6 | 6 | 6 | 6 | 37
  Male | 8 | 8 | 8 | 8 | 8 | 8 | 48

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Plasma Concentration
Time Frame: before OPC dosing, and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-OPC dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- BIA 9-1067 5 mg CM: BIA 9-1067 5 mg CM CM - clinical micronized
- BIA 9-1067 5 mg TBM: BIA 9-1067 5 mg TBM TBM - to-be-marketed
- BIA 9-1067 25 mg CM: BIA 9-1067 25 mg CM CM - clinical micronized
- BIA 9-1067 25 mg TBM: BIA 9-1067 25 mg TBM TBM - to-be-marketed
- BIA 9-1067 50 mg CM: BIA 9-1067 50 mg CM CM - clinical micronized
- BIA 9-1067 50 mg TBM: BIA 9-1067 50 mg TBM TBM - to-be-marketed
Arm/Group | BIA 9-1067 5 mg CM | BIA 9-1067 5 mg TBM | BIA 9-1067 25 mg CM | BIA 9-1067 25 mg TBM | BIA 9-1067 50 mg CM | BIA 9-1067 50 mg TBM
Number analyzed (Participants) | 29 | 28 | 28 | 28 | 28 | 28
ng/mL | 107.3 (55.7) | 95.5 (37.8) | 424.5 (155.7) | 471.0 (206.9) | 756.2 (302.4) | 802.9 (363.0)

2. Secondary Outcome: AUC0-t - Area Under the Plasma Concentration-time Curve for BIA 9-1067
Description: Area Under the plasma concentration-time Curve from time 0 to the time of last quantifiable concentration
Time Frame: before OPC dosing, and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-OPC dose
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | BIA 9-1067 5 mg CM | BIA 9-1067 5 mg TBM | BIA 9-1067 25 mg CM | BIA 9-1067 25 mg TBM | BIA 9-1067 50 mg CM | BIA 9-1067 50 mg TBM
Number analyzed (Participants) | 29 | 28 | 28 | 28 | 28 | 28
ng.h/mL | 196.8 (128.5) | 197.7 (89.7) | 1137 (413.8) | 1270 (515.5) | 2043 (1032) | 2161 (1110)

3. Secondary Outcome: Tmax - Time of Occurrence of Cmax
Time Frame: before OPC dosing, and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-OPC dose
Measure: Median (Full Range); unit: hours
Arm/Group | BIA 9-1067 5 mg CM | BIA 9-1067 5 mg TBM | BIA 9-1067 25 mg CM | BIA 9-1067 25 mg TBM | BIA 9-1067 50 mg CM | BIA 9-1067 50 mg TBM
Number analyzed (Participants) | 29 | 28 | 28 | 28 | 28 | 28
hours | 2.00 [0.50 to 4.00] | 1.00 [0.50 to 4.00] | 2.00 [0.50 to 4.00] | 2.00 [0.50 to 4.00] | 2.00 [1.00 to 4.00] | 2.00 [1.00 to 4.00]

ADVERSE EVENTS:
Arm/Group | BIA 9-1067 5 mg CM | BIA 9-1067 5 mg TBM | BIA 9-1067 25 mg CM | BIA 9-1067 25 mg TBM | BIA 9-1067 50 mg CM | BIA 9-1067 50 mg TBM
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28 | 1/28 | 0/28 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 1/29 | 3/28 | 6/28 | 3/28 | 1/28 | 3/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 9-1067 5 mg CM (N=29) | BIA 9-1067 5 mg TBM (N=28) | BIA 9-1067 25 mg CM (N=28) | BIA 9-1067 25 mg TBM (N=28) | BIA 9-1067 50 mg CM (N=28) | BIA 9-1067 50 mg TBM (N=28)
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 9-1067 5 mg CM (N=29) | BIA 9-1067 5 mg TBM (N=28) | BIA 9-1067 25 mg CM (N=28) | BIA 9-1067 25 mg TBM (N=28) | BIA 9-1067 50 mg CM (N=28) | BIA 9-1067 50 mg TBM (N=28)
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 2 | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other